CLINICAL TRIAL: NCT00126984
Title: A Phase II, Open (Partially Double-blind), Randomized, Controlled Dose-range Study to Evaluate the Immunogenicity, Reactogenicity and Safety of Investigational Vaccination Regimens Versus MENINGITEC™ or MENCEVAX™ ACWY When Given as One Dose to Children Aged 12 to 14 Months and 3 to 5 Years Old
Brief Title: Study in Children to Evaluate the Immunogenicity and Safety of 4 Formulations of GSK Bio MenACWY-TT Conjugate Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 104703 (Primary study); 104704 (Other: GSK)
Record Dates: First submitted 2005-08-04; First posted 2005-08-05 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-10

CONDITIONS: Infections, Meningococcal
Keywords: Safety; Reactogenicity; Immunogenicity; Meningococcal vaccine; Dose selection; Conjugate vaccine
MeSH Terms: conditions — Meningococcal Infections | interventions — Vaccines; PsACWY vaccine

ARMS (5):
- Group A (Experimental): Subjects of 12-14 months of age or 3-5 years of age who will receive formulation A
  Interventions: Biological: Conjugated meningococcal ACWY-TT (vaccine); Biological: DTPa/Hib containing vaccine
- Group B (Experimental): Subjects of 12-14 months of age or 3-5 years of age who will receive formulation B
  Interventions: Biological: Conjugated meningococcal ACWY-TT (vaccine); Biological: DTPa/Hib containing vaccine
- Group C (Experimental): Subjects of 12-14 months of age or 3-5 years of age who will receive formulation C
  Interventions: Biological: Conjugated meningococcal ACWY-TT (vaccine); Biological: DTPa/Hib containing vaccine; Biological: Mencevax ACWY
- Group D (Experimental): Subjects of 12-14 months of age or 3-5 years of age who will receive formulation D
  Interventions: Biological: Conjugated meningococcal ACWY-TT (vaccine); Biological: DTPa/Hib containing vaccine
- Group E (Active Comparator): Subjects of 12-14 months of age who will receive Meningitec and subjects of 3-5 years of age who will receive Mencevax ACWY.
  Interventions: Biological: DTPa/Hib containing vaccine; Biological: Meningitec; Biological: Mencevax ACWY

INTERVENTIONS:
Biological: Conjugated meningococcal ACWY-TT (vaccine) — One intramuscular dose during the primary vaccination
  Arms: Group A; Group B; Group C; Group D
Biological: DTPa/Hib containing vaccine — One intramuscular dose during the primary vaccination study in subjects of 12-14 months of age
Biological: Meningitec — One intramuscular dose during the primary vaccination study in subjects of 12-14 months of age
  Arms: Group E
Biological: Mencevax ACWY — One subcutaneous dose during the primary vaccination study in subjects of 3-5 years of age (group E) and subcutaneous administration of 1/5 dose during the booster vaccination study in subjects of 12-14 months of age (group C, group E)
  Arms: Group C; Group E

SUMMARY:
The purpose of this study is to evaluate the immunogenicity, safety and reactogenicity of one dose of four different formulations of the MenACWY conjugate vaccine when given to healthy children aged 12 14 months and 3 5 years. The selection of the best formulation will be based on data obtained up to one month after the vaccine dose. The Protocol Posting has been updated in order to comply with the FDA Amendment Act, September 2007.

DETAILED DESCRIPTION:
The study will enrol subjects of 12 to 14 months of age and subjects of 3 to 5 years of age. Meningitec™ or Mencevax™ ACWY vaccine will serve as active control. The study will be conducted in two stages: The primary vaccination phase (Study Stage 1) of the study will include all subjects; the second (booster/persistence) phase of the study (Study Stage 2) will include subjects in the active control groups and in the group which was primed with the selected MenACWY formulation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parents/guardians can and will comply with the requirements of the protocol
* A male or female between, and including, 12 and 14 months or 3 and 5 years of age at the time of the first vaccination
* Written informed consent obtained from the parent or guardian of the subject.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study
* Previously completed routine childhood vaccinations to the best of his/her parents'/guardians' knowledge. For pertussis vaccination, the children aged 12-14 months should have been vaccinated with an acellular pertussis vaccine.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Planned administration/ administration of a vaccine not foreseen by the study protocol within one month of the first dose of vaccine and up to one month after administration of each study vaccine dose with the exception of oral polio vaccine.
* Previous vaccination against meningococcal serogroup A, C, W-135 or Y disease.
* Administration of a H. influenzae type b, diphtheria or tetanus vaccine within 3 months before the first dose of vaccine.
* For subjects aged 12-14 months at enrolment, a DTPa/Hib containing booster vaccination, in the second year of life: these booster vaccines will be given at Visit 2.
* History of meningococcal serogroup A, C, W-135 or Y disease.
* Known exposure to meningococcal serogroup A, C, W-135 or Y disease within the previous year.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection.
* A family history of congenital or hereditary immunodeficiency.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Major congenital defects or serious chronic illness.
* History of any neurologic disorders or seizures.
* Acute disease at the time of enrolment.
* Administration of immunoglobulins and/or any blood products within the three months preceding the first dose of study vaccine or planned administration during the study period.

Ages: 12 Months to 14 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 508 (Actual)
Dates: Start 2005-07; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Percentage of meningococcal rSBA responders, in all subjects | One month after the first vaccine dose

SECONDARY OUTCOMES:
Meningococcal rSBA titres | Prior to & 1 month after the 1st dose in all subjects and 15 months after priming in all subjects of groups C and E and one month after administration of the Mencevax ACWY booster dose in all subjects who received the booster dose
Anti-meningococcal polysaccharide concentrations | Prior to & 1 month after the 1st dose in all subjects and 15 months after priming in all subjects of groups C and E and one month after administration of the Mencevax ACWY booster dose in all subjects who received the booster dose
Anti-tetanus toxoid seropositivity and antibody concentrations | Prior to and one month after administration of the first vaccine dose, in all subjects
Meningococcal hSBA titers | Prior to & 1 month after the 1st dose and 15 months after priming in all subjects of groups C and E and one month after administration of the Mencevax ACWY booster dose in all subjects who received the booster dose
Occurrence of local and general solicited adverse events | During the 8-day follow-up period following the administration of each vaccine dose.
Occurrence of unsolicited adverse events | During the 31-day follow-up period following the administration of each vaccine dose.
Occurrence of any serious adverse events | Throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (33):
- Austria (5):
  - GSK Investigational Site, Güssing
  - GSK Investigational Site, Neufeld/Leitha
  - GSK Investigational Site, Salzburg
  - GSK Investigational Site, Villach
  - GSK Investigational Site, Wels
- Germany (28):
  - GSK Investigational Site, Bietigheim-Bissingen, Baden-Wurttemberg
  - GSK Investigational Site, Bretten, Baden-Wurttemberg
  - GSK Investigational Site, Eppelheim, Baden-Wurttemberg
  - GSK Investigational Site, Ludwigsburg, Baden-Wurttemberg
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Oberstenfeld, Baden-Wurttemberg
  - GSK Investigational Site, Bindlach, Bavaria
  - GSK Investigational Site, Bobingen, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Nördlingen, Bavaria
  - GSK Investigational Site, Nuremberg, Bavaria
  - GSK Investigational Site, Olching, Bavaria
  - GSK Investigational Site, Tegernsee, Bavaria
  - GSK Investigational Site, Tutzing, Bavaria
  - GSK Investigational Site, Weilheim, Bavaria
  - GSK Investigational Site, Bodenheim, Rhineland-Palatinate
  - GSK Investigational Site, Gerolstein, Rhineland-Palatinate
  - GSK Investigational Site, Ludwigshafen am Rhein, Rhineland-Palatinate
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Trier, Rhineland-Palatinate
  - GSK Investigational Site, Worms, Rhineland-Palatinate
  - GSK Investigational Site, Döbeln, Saxony
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Stollberg, Saxony
  - GSK Investigational Site, Berlin, State of Berlin
  - GSK Investigational Site, Bad Lobenstein, Thuringia
  - GSK Investigational Site, Weimar, Thuringia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Knuf M, Kieninger-Baum D, Habermehl P, Muttonen P, Maurer H, Vink P, Poolman J, Boutriau D. A dose-range study assessing immunogenicity and safety of one dose of a new candidate meningococcal serogroups A, C, W-135, Y tetanus toxoid conjugate (MenACWY-TT) vaccine administered in the second year of life and in young children. Vaccine. 2010 Jan 8;28(3):744-53. doi: 10.1016/j.vaccine.2009.10.064. Epub 2009 Nov 1. PMID 19887137
- [Background] Knuf M, Baine Y, Bianco V, Boutriau D, Miller JM. Antibody persistence and immune memory 15 months after priming with an investigational tetravalent meningococcal tetanus toxoid conjugate vaccine (MenACWY-TT) in toddlers and young children. Hum Vaccin Immunother. 2012 Jul;8(7):866-72. doi: 10.4161/hv.20229. Epub 2012 Apr 9. PMID 22485049
- [Background] Knuf M et al. Antibody persistence and immune memory 15 months after meningococcal tetravalent tetanus toxoid conjugate (ACWY-TT) vaccine in toddlers and 3-5 year-olds. Abstract presented at the 27th annual ESPID meeting, Brussels, Belgium, 9-13 June 2009.
- [Background] Prieler et al. Immunogenicity of 1 dose of a candidate meningococcal tetravalent tetanus toxoid conjugate (MenACWY-TT) vaccine in 12-14 month and 3-5 year olds. Abstract presented at the 47th Annual Meeting of Interscience Conference on Antimicrobial Agents and Chemotherapy (ICAAC). Chicago, IL, 17-20 September 2007.
- [Background] Prieler et al. Immunogenicity of 1-dose of a new meningococcal serogroups A, C, W-135, Y tetanus toxoid conjugate (MenACWY-TT) vaccine in children 12-14 months and 3-5 years old. Abstract presented at the 9th Meeting of The European Monitoring Group on Meningococci (EMGM). Rome, Italy, 30 May-1 June 2007.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 104703 (Primary study) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 104703 (Primary study) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 104703 (Primary study) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 104703 (Primary study) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 104703 (Primary study) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register. The results of this study 104703 are summarised with study 104704 on the GSK Clinical Study Register.
- Available data/document: Dataset Specification: 104703 (Primary study) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register